CLINICAL TRIAL: NCT01462188
Title: Immediate Versus Delayed Stenting in Patients With ST-Elevation Myocardial Infarction Undergoing Mechanical Intervention
Brief Title: Optimizing Infarct Size by Transforming Emergent Stenting Into an Elective Procedure Study
Acronym: OPTIMASTRATEGY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marco Valgimigli (Other)
Responsible Party: Sponsor-Investigator, Marco Valgimigli, Head of the Catheterization laboratory, Università degli Studi di Ferrara
Organization: Università degli Studi di Ferrara (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRAPS-09-I
Record Dates: First submitted 2011-10-24; First posted 2011-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Myocardial Infarction
Keywords: ST-segment elevation myocardial infarction; Primary angioplasty; stent
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate stenting (Active Comparator): Patients being randomized to the immediate stenting arm will be managed according to the guidelines. Irrespective of TIMI flow at presentation, investigators will be requested to thrombus aspirate immediately after successful wiring of the culprit vessel followed by direct stenting. In cases where insertion of thrombus removal catheter and/or direct stenting is not successful, balloon angioplasty will be allowed.
  Interventions: Procedure: Immediate stenting
- Delayed stenting (Experimental): Patients being randomized to the delayed/staged stenting arm will be managed with the aim to obtain stable TIMI 3 flow with no considerations given at the percentage of residual stenosis at the culprit lesion.
  In patients presenting with TIMI 3 flow, investigators will be left free to wire the vessel and proceed to thrombus aspiration to decrease thrombus burden in the culprit lesion or to leave the vessel untreated at the time of index PCI. Patients presenting with suboptimal TIMI flow (i.e. less than 3), investigators are required to wire the vessel and thrombus aspirate. If stable (persisting for at least 5 minutes) TIMI 3 flow is obtained, investigators are requested to stop the procedure. The goal is to achieve s table TIMI 3 flow with no considerations given to the percentage of residual stenosis. Stenting in this arm will be allowed only on a bail-out strategy.
  Interventions: Procedure: Delayed stenting

INTERVENTIONS:
Procedure: Immediate stenting — Primary coronary stenting
  Arms: Immediate stenting
Procedure: Delayed stenting — Coronary stenting 3 to 7 days after having reopened the vessel in the acute phase
  Arms: Delayed stenting

SUMMARY:
The goal of primary PCI is to restore anterograde myocardial flow. Stenting a largely thrombotic lesion may determine distal embolisation of thrombotic material therefore deteriorating myocardial perfusion.

DETAILED DESCRIPTION:
In the setting of largely thrombotic lesions such as those treated in the context of primary PCI, stenting often results in distal micro and macro-embolisation which hampers coronary flow and microvascular recovery. Interestingly in some of these studies comparing BMS versus balloon angioplasty an early hazard associated to the use of stent has been reported.

Thus, investigators hypothesize in this protocol that refraining from stenting during the acute phase of ST segment myocardial infarction is safe and associated to improved myocardial recovery as compared to acute stenting.

ELIGIBILITY:
Inclusion Criteria:

* chest pain for >30 min with ST-segment elevation of one mm or more in 2 or more contiguous ECG leads or with presumably new left bundle-branch block
* admission either within 12 h of symptom onset or between 12 and 24 h with evidence of continuing ischaemia

Exclusion Criteria:

* the exclusion criteria will include history of bleeding diathesis or documented allergy/intolerance or contraindication to clopidogrel or ticlopidine or prasugrel
* inability to assume an oral P2Y12 receptor blocker on a consecutive daily basis for a minimum of 6 months, or to heparin or aspirin
* uncontrolled hypertension (systolic or diastolic arterial pressure >180 mmHg or 120, respectively, despite medical therapy)
* limited life expectancy, e.g. neoplasms, others
* inability to obtain informed consent
* pregnancy
* patients were not enrolled if they were clinically unstable, presented with severe arrhythmia, or had known contraindications to CMR (claustrophobia, pacemakers, or implantable defibrillator devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Myocardial blush grade (MBG) equal or greater than 2 | post-procedure
  The MBG will be estimated visually by 2 experienced observers, as previously described.

SECONDARY OUTCOMES:
ST segment elevation resolution | 30 minutes after the procedure
  Cumulative ST segment elevation in all leads will be quantified before and after the procedure and expressed as percentage
ST segment elevation Resolution | 90 minutes after the procedure
infarct size | 5 days
  Infarct size will be quantified by MRI
Infarct size | 6 months
  Infarct size will be quantified by MRI
microvascular obstruction | 5 days
  microvascular obstruction will be quantified by MRI
microvascular obstruction | 6 months
  microvascular obstruction will be quantified by MRI
Mortality | 6 months
  overall and cardiac mortality will be assessed up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Cardiologia, Ferrara, Emilia-Romagna, Italy